CLINICAL TRIAL: NCT01320904
Title: Neuromuscular Electrical Stimulation (NMES) on Knee Osteoarthritis(OA): an Equivalence Randomized Clinical Trial
Brief Title: Exercise and Muscle Stimulation in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Luterana do Brasil (Other)
Responsible Party: Marcelo Baptista Dohnert, Universidade Luterana do Brasil
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MBD 275767
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Osteoarthritis, Knee; Self Stimulation; Exercise Addiction
Keywords: Closed Kinetic Chain; NMES; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Self Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed Kinetic Chain and NMES placebo (Placebo Comparator): During the stimulation period the patient remained in a mini-squat position at thirty degrees and returned to zero degrees during the decay period. During the electrical stimulation off period, the patient spontaneously performed another mini-squat at 30 degrees without electrical stimulation. The patients in the CKC + NMES placebo group simulated the same work applied to the NMES group. Notably, this group was also connected to the electrodes, but the equipment was set at a stimulus intensity of zero.
  We used a 10-channel electrical stimulation device with a 2500-Hz carrier frequency. We used four channels in the synchronous mode, with surface electrodes that were simultaneously fixed at the motor points of the quadriceps and hamstrings.
  Interventions: Procedure: NMES
- Closed Kinetic Chain Group (Other): During the stimulation period, i.e., the on time, the patient remained in a mini-squat position at thirty degrees and returned to zero degrees during the decay period. During the electrical stimulation off period, the patient spontaneously performed another mini-squat at 30 degrees without electrical stimulation. The patients in the CKC + NMES placebo group simulated the same work applied to the NMES group. Notably, this group was also connected to the electrodes, but the equipment was set at a stimulus intensity of zero.
  Interventions: Procedure: Closed Kinetic Chain

INTERVENTIONS:
Procedure: NMES — We used a electrical stimulation device with a 2500-Hz carrier frequency. We used four channels in the synchronous mode, with surface electrodes that were simultaneously fixed at the motor points of the quadriceps and hamstrings. Initially, a warm-up protocol that was five minutes long was used at a stimulation frequency of 40 Hz to activate the slow fibers. These fibers activated with a four-second-contraction time (on), a four-second-stimulus rise time, a four-second-stimulation decay time and a 12-second relaxation time (off).
  We then increased the frequency to 70 Hz to activate the fast fibers for an additional 10 minutes using the parameters described above, and finally, the frequency was increase to 150 Hz for 10 minutes to achieve maximal muscle potentiation.
  Other Names: 10-channel NEURODYN electrical stimulation IBRAMED
  Arms: Closed Kinetic Chain and NMES placebo
Procedure: Closed Kinetic Chain — During the stimulation period, i.e., the on time, the patient remained in a mini-squat position at thirty degrees and returned to zero degrees during the decay period. During the electrical stimulation off period, the patient spontaneously performed another mini-squat at 30 degrees without electrical stimulation. The patients in the CKC + NMES placebo group simulated the same work applied to the NMES group. Notably, this group was also connected to the electrodes, but the equipment was set at a stimulus intensity of zero.
  Other Names: Closed Kinetic Chain exercises
  Arms: Closed Kinetic Chain Group

SUMMARY:
Objective: To evaluate the effectiveness of neuromuscular electrical stimulation (NMES) combined with closed kinetic chain (CKC) exercises in patients with knee OA.

DETAILED DESCRIPTION:
Abstract:

Introduction: Osteoarthritis (OA) is a degenerative and debilitating change that affects the synovial joints.

Objective: To evaluate the effectiveness of neuromuscular electrical stimulation (NMES) combined with closed kinetic chain (CKC) exercises in patients with knee OA.

Methods: Nineteen patients with knee OA were enrolled and randomized into two groups: group I was treated with CKC + NMES, and group II was treated with CKC + NMES placebo. Both groups underwent 20 sessions of mini-squat exercises at 30 degrees of knee flexion that were associated with and interspersed with NMES for 5 minutes at a frequency of 40 hertz (Hz), 10 minutes at 70 Hz and an addition 10 minutes at 150 Hz, for a total of 25 minutes. The data were analyzed using SPSS (Statistical Package for the Social Sciences) version 17.0. Data were expressed as a frequency, mean and standard deviation and were statistically analyzed using a one-way analysis of variance (ANOVA) for repeated measurements followed by Bonferroni's post-hoc test. The investigators also used an unpaired Student's t-test and Kruskal-Wallis and Wilcoxon tests with a level of significance of P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with grade I or grade II knee OA (based on the Kellgren-Lawrence classification;
* which was diagnosed by a medical traumatologist;
* radiographic changes that demonstrated a reduced joint space in at least one of the compartments of the knee;
* subchondral bone sclerosis;
* consent to participate in the study

Exclusion Criteria:

* patients who had grade III and grade IV knee OA (based on the Kellgren-Lawrence classification);
* who were involved in another rehabilitation program outside the center;
* who presented with clinical symptoms that would prevent them from participating in the exercises;
* who had heart disease;
* cardiac pacemakers;
* periarticular metal implants;
* who experienced changes in sensitivity;
* who had a previous history of knee injury (meniscus, ligaments, sprains);
* who had uncontrolled diabetes;
* neurological disorders with cognitive impairments;
* rheumatic diseases;
* history of knee trauma in the last six months;
* prior knee surgery;
* three consecutive unexcused absences.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the flexibility of the posterior chain muscles | 6 months
  We only observed a significant improvement in the flexibility of the posterior muscle chain for the CKC + NMES group during the initial evaluation compared to the partial evaluation (p=0.012), the partial evaluation compared to the final evaluation (p=0.035) and the initial evaluation compared to the final evaluation (p=0.008). Regarding the scale that was used to classify the level of flexibility, 10% of the subjects in the CKC + NMES group were initially classified as good/excellent. At the end of the protocol, 60% of the subjects were classified as good/excellent (p=0.015)

SECONDARY OUTCOMES:
Evaluation of hamstring and quadriceps muscle strength | 6 months
  A significant improvement in muscle strength was only observed in the group treated with CKC + NMES. The improvement in quadriceps strength occurred during the first 10 sessions (p=0.001) Muscle strength in the hamstring muscle group responded similarly to the quadriceps muscle group (i.e., a significant improvement in muscle strength was only observed in the CKC + NMES group) in both the initial evaluation compared to the partial evaluation at 10 sessions (p=0.009) and the initial evaluation compared to the final evaluation (p=0.006)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Dohnert, Principal Investigator — Universidade Luterana do Brasil